CLINICAL TRIAL: NCT05337605
Title: Hand Driven Versus Motor Driven Hysteroscopic Tissue Removal System for Polypectomy: Long-term Results
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-11626 BC-11627 BC-11628
Record Dates: First submitted 2022-04-04; First posted 2022-04-20 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Endometrial Polyp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hand driven tissue removal system: Endometrial polyp removed by hysteroscopic hand-driven tissue removal system in a previous study.
- Motor driven tissue removal system: Endometrial polyp removed by hysteroscopic motor-driven tissue removal system in a previous study.

SUMMARY:
In this study, a comparison is made between two types of polyp resection methods (hand driven and motor driven morcellation). More specifically, the effects of the resection on symptoms such as abnormal uterine bleeding, and on the recurrence of polyps.

The aim of the study is to find a superior method in terms of symptom relieve and polyp recurrence so this method can be used in gynaecological practice.

DETAILED DESCRIPTION:
* Rationale: several techniques for hysteroscopic removal of intrauterine polyps exist today. Hysteroscopic morcellation is an effective, fast, and safe method for this. However, the differences between two different systems of hysteroscopic morcellation, motor-driven (Truclear incisor mini device) and hand-driven (Resectr 9fr) morcellation, are still unclear. The REMOvE9 study, in which women with a polyp were randomized between both techniques, is currently investigating the differences in short-term effectiveness between the two techniques.
* Research question/goal: To investigate the long-term results of the effectiveness of a hysteroscopic morcellation of intrauterine polyps. The two systems are compared with each other.
* Study design: This is a prospective cohort study. The patients previously participated in a randomized controlled trial (REMOvE9) and will now be contacted again for the completion of a one-time questionnaire. The study has an observational design.
* Study population: Women with a history of endometrial polyp that was previously removed via hysteroscopic morcellation in the REMOvE9 study.
* Primary and secondary endpoints: The primary endpoint is the risk of recurrence of abnormal uterine bleeding at post-surgery follow-up. Secondary endpoints include recurrence of other symptoms, time to recurrence, symptom relief, onset of new symptoms, onset of new polyp, satisfaction with regards to symptoms, satisfaction with regards to the treatment in general, need for additional treatments for blood loss and occurrence of pregnancy (in subfertility group).

ELIGIBILITY:
Inclusion Criteria:

* participation in earlier study

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women treated for endometrial polyps in earlier study
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Rate of recurrence of abnormal uterine blood loss (+ cause, treatment) | 1 to 4 years
  Patient reported outcome by means of a questionnaire (yes/no, specify)

SECONDARY OUTCOMES:
Rate of recurrence of other symptoms (abdominal pain, infections, back pain, other..) (+ cause, treatment) | 1 to 4 years
  Patient reported outcome by means of a questionnaire (yes/no, specify)
Recurrence interval (time to recurrence of endometrial polyp) | 1 to 4years
  Patient reported outcome by means of a questionnaire (when did blood loss occur / when was polyp identified)
Number of patients with symptom relief after initial intervention (abdominal pain, abnormal uterine blood loss, other...) | 1 to 4years
  Patient reported outcome by means of a questionnaire
Rate of occurrence of new symptoms after initial intervention (abdominal pain, abnormal uterine blood loss, infections, other...) (+ cause, treatment) | 1 to 4years
  Patient reported outcome by means of a questionnaire (yes/no, specify)
Rate of occurrence of new polyps (+ cause, treatment) | 1 to 4years
  Patient reported outcome by means of a questionnaire (yes/no, specify)
Satisfaction score in regard to symptoms (abdominal pain, abnormal uterine blood loss, other...) | 1 to 4years
  Patient reported outcome by means of a questionnaire on a scale from 0 (bad) to 5 (great)
General satisfaction score in regard to initial treatment | 1 to 4years
  Patient reported outcome by means of a questionnaire on a scale from 0 (bad) to 5 (great)
Rate of need for additional treatment | 1 to 4years
  Patient reported outcome by means of a questionnaire (yes/no, specify)
Chance of pregnancy after treatment | 1 to 4 years
  Only applicable for women with fertility problems, Patient reported outcome by means of a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Tjalina Hamerlynck, Md, Phd, Principal Investigator — University Hospital, Ghent
Locations (1):
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Van Geyte M, de Frenne A, Weyers B, Weyers S, van Vliet H, Hamerlynck T, van Wessel S. Manually driven versus motor driven hysteroscopic tissue removal system for polypectomy: Long-term results. Eur J Obstet Gynecol Reprod Biol. 2024 May;296:270-274. doi: 10.1016/j.ejogrb.2024.03.013. Epub 2024 Mar 12. PMID 38492506